CLINICAL TRIAL: NCT00217919
Title: Reducing Risk Factors in Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 296; R01HL073912 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Health-Counselor Mediated Telephone Counseling Intervention
  Interventions: Behavioral: Health-Counselor Mediated Telephone Counseling Intervention
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Health-Counselor Mediated Telephone Counseling Intervention — A trained health counselor will conduct the TC sessions, which will occur every 6 weeks (total 8 calls). We expect the initial call to last 30 minutes, with subsequent calls lasting 20 minutes. Our intervention for our primary outcome of LDL-C lowering is expected to take most of this time. We will spend approximately 5 minutes addressing physical activity at the end of each session, using methods similar to those in our pilot TC study.
  We will use patient-centered counseling to promote adherence to lipid-lowering medication and LDL-C lowering diet. The intervention will also activate patients to discuss initiation or dose increase of lipid-lowering drugs with their physicians. While the focus of our intervention will be on LDL-C lowering, the TC intervention will also devote approximately 5 minutes of the typical 20 minute call to increasing physical activity.
  Arms: 1

SUMMARY:
The purpose of this study is to compare a health-counselor mediated telephone counseling intervention to usual care to reduce low density lipoprotein cholesterol (LDL-C) levels in patients with peripheral arterial disease (PAD).

DETAILED DESCRIPTION:
BACKGROUND:

Patients with PAD have a 3- to 4-fold higher risk of cardiovascular morbidity and mortality compared to patients without PAD. Risk of future cardiovascular events is comparable between patients with PAD and coronary artery disease (CAD). While improved atherosclerotic risk factor treatment has reduced cardiovascular morbidity and mortality in patients with CAD, such treatment in patients with PAD remains suboptimal. Intensity of cholesterol-lowering therapy, specifically, is significantly poorer in patients with PAD as compared to CAD. Data show that fully 69 percent of patients with PAD from a non-invasive vascular laboratory in Chicago did not have the recommended LDL-C level of less than 100 mg/dl. Our data from a national survey indicate that physicians believe atherosclerotic risk factor treatment is less important for patients with PAD than for patients with CAD. Our data also show that many patients with PAD are unaware of their increased risk of cardiovascular events and under-appreciate the importance of risk factor treatment in PAD. These findings likely contribute to risk factor under-treatment in patients with PAD. Clinical trials such as this are needed to demonstrate whether PAD risk factors can be reduced. If effective, this clinical trial will also encourage clinicians to adopt the proven intervention to lower cardiovascular risks in patients with PAD

DESIGN NARRATIVE:

This randomized, controlled clinical trial will test the ability of a health-counselor mediated telephone counseling intervention as compared to usual care to reduce LDL-C levels in patients with PAD. The study involves patients with PAD who have LDL-C levels greater than 100 mg/dl at baseline identified from non-invasive vascular laboratories in Chicago, IL and Worcester, MA. For their primary specific aim, the investigators hypothesize that subjects randomized to the intervention condition will achieve a reduction in LDL-C of at least 11.1 mg/dl greater than the reduction in LDL-C for subjects randomized to the usual care condition at 12-month follow-up. In their secondary aim, they will determine whether the telephone counseling intervention increases the proportion of PAD patients with LDL-C less than 100 mg/dl as compared to the usual care condition at 12-month follow-up. To identify the mediators of the intervention, in their exploratory aims they will determine whether patients in the intervention condition achieve greater increases (improvement) in specific behavioral and knowledge and attitude mediators that will be targeted by the intervention, as compared to patients in the usual care condition.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy greater than 1 year
* Has a telephone
* English-speaking
* Willing to use acceptable methods of contraception
* Have a primary care physician

Exclusion Criteria:

* Currently undergoing cancer treatment or plans to begin treatment
* Psychiatric illness or cognitive impairment
* Intolerance to two or more cholesterol-lowering drugs
* Plans to move out of the area within one year of study entry
* Wheel-chair bound or unable to walk outside of home
* Below- or above-knee amputation
* Unstable angina
* Current foot ulcers
* LDL-C less than 70 mg/dl at baseline
* Debilitating chronic obstructive lung disease
* Major surgery within 3 months prior to study entry or plans to undergo major surgery within 1 year of study entry
* Current participation in another clinical trial. A six month period will be required after completing another clinical trial before an individual can become eligible for the current trial.
* Ischemic rest pain
* Pregnancy or plan to become pregnant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2006-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
LDL-C levels | Measured at baseline and Month 12
LDL-C lowering knowledge, attitude, and behavior | Measured at baseline and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Mary McDermott, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts

REFERENCES:
- [Derived] Pagoto SL, McDermott MM, Reed G, Greenland P, Mazor KM, Ockene JK, Whited M, Schneider K, Appelhans B, Leung K, Merriam P, Ockene I. Can attention control conditions have detrimental effects on behavioral medicine randomized trials? Psychosom Med. 2013 Feb;75(2):137-43. doi: 10.1097/PSY.0b013e3182765dd2. Epub 2012 Nov 28. PMID 23197844
- [Derived] McDermott MM, Greenland P, Reed G, Mazor KM, Merriam PA, Graff R, Tao H, Pagoto S, Manheim L, Kibbe MR, Ockene IS. Gender differences in cholesterol-lowering medication prescribing in peripheral artery disease. Vasc Med. 2011 Dec;16(6):428-35. doi: 10.1177/1358863X11425879. PMID 22128042
- [Derived] McDermott MM, Reed G, Greenland P, Mazor KM, Pagoto S, Ockene JK, Graff R, Merriam PA, Leung K, Manheim L, Kibbe MR, Olendzki B, Pearce WH, Ockene IS. Activating peripheral arterial disease patients to reduce cholesterol: a randomized trial. Am J Med. 2011 Jun;124(6):557-65. doi: 10.1016/j.amjmed.2010.11.032. PMID 21605733
- [Derived] McDermott MM, Mazor KM, Reed G, Pagoto S, Graff R, Merriam P, Kibbe M, Greenland P, Ockene J, Olendzki B, Huimin Tao, Ockene I. Attitudes and behavior of peripheral arterial disease patients toward influencing their physician's prescription of cholesterol-lowering medication. Vasc Med. 2010 Apr;15(2):83-90. doi: 10.1177/1358863X09353653. Epub 2010 Jan 29. PMID 20118170